CLINICAL TRIAL: NCT03747133
Title: Phase II Study: Stereotactic Ablative Radiotherapy for Renal Tumors
Brief Title: SABR for Renal Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-5481
Record Dates: First submitted 2018-11-01; First posted 2018-11-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Renal Tumor
Keywords: Stereotactic Body Radiation Therapy; SABR; Radiation Therapy; Renal Cell Carcinoma; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Ablative Radiotherapy (Experimental): Adult patients with Kidney mass (either primary or metastasis) amenable to SABR
  Interventions: Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy — Stereotactic Ablative Radiotherapy to renal tumors with a dose of 27.5-40 Gy in 5 fractions.

SUMMARY:
Renal Cell Carcinoma (RCC) is the most common type of kidney cancer. The usual treatment for this type of cancer is surgery. Considering the most common patients are an average age of 65 and some are not suitable candiates for surgery, there is great interest in non-surgical alternatives for kidney cancer treatments. This study will investigate the use of Stereotactic Ablative Radiosurgery (SABR) for renal tumors. SABR is a non-invasive alternative, which involves delivery of high doses of radiation to the target, while minimizing the risk of injury to the surrounding organs. Patients will be seen before and end of treatmetn and will be followed at 4 month intervals for up to 2 years. During the follow ups, patients will be asked to complete a quality of life questionnaire and will have standard of care imaging.

ELIGIBILITY:
Inclusion Criteria:

* Solid Kidney Mass (primary RCC or metastasis) amenable to SABR ≤6cm
* Histological or radiological diagnosis of renal tumor
* Inoperable: High risk for surgery or declined surgery
* ECOG performance status of 0-3

Exclusion Criteria:

* ≥5 active metastases
* Sysstemic therapy (except endocrine therapy) wthin 6 days prior to SABR
* Prior abdominal radiotherapy with fields overlap resulting in excessive doses to the involved kidney
* Patients with end stage renal failure > 4(KDOQI guidelines)
* Familial Syndrome: Von Hippel-Lindau disease, Polycystic Kidney Disease, Hereditary Papillary RCC or Tuber Sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the radiation induced renal impairments in patients receiving SABR. | 2 years
  The prevalence of nephron toxicity in patients treated with SABR, measured by the change in Glomerular Filtration Rate (GFR) every 4 months over 2 years.

SECONDARY OUTCOMES:
Chronic Kidney Disease Stage Progression | 2 years
  Chronic kidney disease stage progression after SABR, assessed by the Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines
2-year Local recurrence rate | 2 years
  2 year local recurrence rate of kidney tumors treated with SABR, measured by assessing the change of irradiated kidney function on functional imaging.
Patient Reported Outcomes | 2 years
  The change in quality of life of patients treated with SABR, assessed through the use of NCCN FKSI-19 questionnaire.
Incidence of acute and late toxicities | 2 years
  The incidence of acute (≤3 months) and late complication of interest (GI or GU complications, high blood pressure and adrenal insufficiency) as assessed by CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McPartlin, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (2):
- Canada (2):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Glicksman RM, Winter J, McPartlin A, Santiago AT, Wang K, Bernstein J, Dang J, Tsui G, Chung P, Mesci A, Gutierrez Valencia E, Raman S, Berlin A, Catton C, Bayley A, Warde P, Krishna S, Finelli A, Hamilton RJ, Pace KT, Kitchlu A, Helou J. Stereotactic Body Radiation Therapy for Renal Tumors: A Prospective Phase 2 Clinical Trial. Int J Radiat Oncol Biol Phys. 2025 Nov 23:S0360-3016(25)06480-6. doi: 10.1016/j.ijrobp.2025.11.005. Online ahead of print. PMID 41290048